CLINICAL TRIAL: NCT00257634
Title: Dexamethasone Delivery for Treatment of Lateral Epicondylitis (IRB #3260)
Brief Title: Randomized Trial of Iontophoresis Versus Injection of Corticosteroids for Lateral Epicondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Birch Point Medical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HFHS-3260
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Lateral Epicondylitis; Work Related Injury
Keywords: lateral epicondylitis; iontophoresis; dexamethasone
MeSH Terms: conditions — Tennis Elbow

INTERVENTIONS:
Drug: dexamethasone to injury site

SUMMARY:
The purpose of this project is to compare different treatment options for lateral epicondylitis. Lateral epicondylitis is a pain condition involving extensor muscles fo the forearm originating from the lateral epicondyle. Controversy exists regarding the method of delivering pain relief so that conditioning and strengthening can be initiated and progress appropriately. Our hypothesis is that the steady even delivery via iontophoresis (compared to injection will provide better pain control and allow physical therapy to progress more effectively.

DETAILED DESCRIPTION:
Therapy is standardized so treatment can begin before enrollment in the study. Patients who decide not to participate will get standard therapy. Therapy is based on the published Indiana Hand Center protocol. Phase 1 is rest, phase 2 is mobility and phase 3 is strengthening. Patients who agree to participate will be randomized to either the injection or iontopatch group after informed consent.

GROUP 1 (injection) Patients seen by physician. Based upon history and physical examination, injection wil be offered. Injection is 10 mg dexamethasone intramuscular. Therapy then is continued per standard protocol. Patient monitored for worsening of symptoms. If the patient worsens, the patient will be placed back into phase 1 and 2 for another 3 weeks then advanced again. Repeat injection will be at discretion of the treating physician. Patients with more than 2 injections wil be disqualified from the study and considered a treatment failure. Patients that injections wil be disqualified from the study and considered a treatment failure. Patients that completed phase 3 will be released from therapy with home management program instructions. Restrictions will be at the discretion of the physician. After 2 failures to progress to phase 3, the patient will be considered a failure of treatment. In the event of relapse after successful completion of therapy, the protocol will be repeated.

GROUP 2 (iontopatch) One volt patch with dexamethasone phosphate will be used.Patient will be treated with one patch every 2 days for a total of 3 patches. Application will be per the Birchpoint Medical Group Iontopatch 80 protocol. The patches will correlate with physical therapy phases 1 and 2. Phase 3 will not begin until the Iontopatch has been off for more than 24 hours. Therapy will progress based on the above protocol. If there is worsening of symptoms, the patient will be placed back to phase 1 and 2 for another 3 weeks and then advanced again. Iontopatches can be repeated if there has been a substantial worsening of symptoms. Patients are eligible for up to 6 patches for the duration of the study. Once the 6 patches have been used, therapy can continue per protocol but without iontopatch and/or injection. Patients that completed phase 3 will be released from therapy. After 2 failures to progress to phase 3, the patient will be considered a failure of treatment. Long term restrictions will be at the discretion of the physician.

Patients will complete a Forearm Pain Questionnaire at the time of enrollment, at completion of therapy and monthly after that for 3 months. This is a standardized published questionnaire specifically designed to identify and track lateral epicondylitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Tenderness at lateral epicondyle,
* No radiographic abnormality at the elbow,
* Mille's Sign positive- pain with elbow extension,
* Forearm pronation,
* Wrist flexion,
* Maudsley Test positive - pain with resisted passive

Exclusion Criteria:

* Pregnancy,
* History of fibromyalgia,
* Elbow surgery,
* Diagnosis of multilevel nerve compression,
* Symptoms of lateral epicondylitis for more than 2 year,
* Bilateral lateral epicondylitis,
* Previous corticosteroid injection in the same elbow,
* Use of systemic steroid medication within the last 6 months,
* Evidence of active infection,
* History of allergic reaction to the study medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-12; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
outcome measurement instrument
grip strength
return to work

SECONDARY OUTCOMES:
cost

CONTACTS AND LOCATIONS:
Overall Officials: aamir siddiqui, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States